CLINICAL TRIAL: NCT01179958
Title: Cognitive Benefits of Aerobic Exercise Across the Age Span
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Principal Investigator, Richard Sloan, Division Chief, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: #6211/7140R; AG030092 (Other: CU)
Record Dates: First submitted 2010-08-10; First posted 2010-08-11 (Estimated); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Cognitive Function
Keywords: cognitive function; fMRI; apoE; inflammatory markers; exercise
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- aerobic training (Experimental): 24 weeks of aerobic training, 4 times/week
  Interventions: Behavioral: aerobic training
- stretching/toning (Placebo Comparator): stretching/toning condition, 24 weeks to parallel the active intervention group
  Interventions: Behavioral: stretching/toning

INTERVENTIONS:
Behavioral: aerobic training — 24 weeks of aerobic training, 4X/week
  Other Names: Training, aerobic
  Arms: aerobic training
Behavioral: stretching/toning — stretches and toning exercises designed to promote flexibility and improved core strength
  Other Names: Exercises, stretches and toning
  Arms: stretching/toning

SUMMARY:
The purpose of this study is to test the hypothesis that aerobic exercise leads improved cognitive function accompanied by increases in gray matter density and changes in functional magnetic resonance imaging (fMRI) patterns of task-related activation.

DETAILED DESCRIPTION:
While animal and human studies indicate cognitive benefits from aerobic exercise across the lifespan, the great majority of controlled exercise studies in humans have been restricted to elderly individuals. Those studies have indicated that enhancing aerobic capacity has a beneficial effect on cognition. One study suggests that this benefit is seen particularly for executive control processes, precisely the processes affected by aging. These improvements have been accompanied by increases in gray matter density and changes in functional magnetic resonance imaging (fMRI) patterns of task-related activation. The goal of the proposed study is to extend the investigation of the beneficial effects of aerobic exercise to younger individuals, and to compare these effects in young and old.

In this application the study team propose to conduct a study in which 270 sedentary but otherwise healthy and cognitively intact individuals in the 20-68 year age range are randomized to two training conditions, aerobic exercise and stretching/toning, to be completed at YMCAs and YMHAs in New York City. Participants will be assessed for aerobic capacity, cognitive task performance, and by structural MRI, resting cerebral blood flow scans (arterial spin labeling) and cognitive activation fMRI studies at study entry and after 6 months of training.

The study also proposes two complementary approaches to investigating the neural correlates of the beneficial effects of aerobic exercise on cognition: 1) imaging -- a combination of structural, metabolic, and cognitive activation fMRI studies to evaluate the neural substrates of the effect of aerobic exercise on cognition will be used. 2) important correlates -- the effects of apolipoprotein E (APOE) genotype, inflammatory markers and cognitive reserve on the cognitive effects of aerobic exercise will be explored.

ELIGIBILITY:
Inclusion Criteria:

1. Age 20-68
2. English-speaking
3. strongly right-handed
4. BMI < 35
5. Pre-menopausal (women only): no oral contraceptive use Post-menopausal: no estrogen replacement therapy
6. sedentary: VO2 max < 41 and 31.6 ml/kg/min for men age 20-40 and 50-68 and < 35.2 and 26.6 ml/kg/min for women age 20-40 and 50-68 respectively
7. participants over age 60 must have ECG within past 3 months

Exclusion Criteria:

1. MRI contraindications (e.g., metallic implants, pacemaker, weight > 350 lbs, waist > 55")
2. Hearing impaired/hearing aids, unable to read newspaper at arm's length with corrective lenses
3. Objective cognitive impairment
4. Ischemic changes, abnormal blood pressure responses, or any significant ectopy during aerobic capacity testing
5. Cardiovascular disease
6. Uncontrolled high blood pressure (systolic blood pressure ≥ 140 mmHg; or diastolic blood pressure ≥ 90 mmHg on two measures)
7. Current or recent (evidence of disease x 5 years) non-skin neoplastic disease or melanoma
8. Active hepatic disease (not a history of hepatitis) or primary renal disease requiring dialysis, primary untreated endocrine diseases, e.g., Cushing's disease or primary hypothalamic failure or insulin dependent diabetes (Type I or II).
9. HIV infection
10. Pregnant or lactating (participation allowed 3 months after ceasing lactation
11. Medications that target CNS (central nervous system, e.g., neuroleptics, anticonvulsants, antidepressants, benzodiazepines) within the last month
12. Women: any selective estrogen receptor modulator or aromatase inhibitor Men: androgen ablation/deprivation hormonal therapies
13. Any history of psychosis or electroconvulsive therapy
14. Psychotic disorder (lifetime)
15. Current or recent (within past 12 months) alcohol or substance abuse or dependence. Recent use (past month) of recreational drugs.
16. Brain disorder such as stroke, tumor, infection, epilepsy, multiple sclerosis, degenerative diseases, head injury, mental retardation
17. Imaged cortical stroke or large subcortical lacunae or infarct or space-occupying lesion (≥ 2 cubic cm). Other findings, e.g., periventricular caps or small white matter hyperintensities, do not result in exclusion
18. Diagnosed learning disability, dyslexia
19. Current or recent (Past 5 years) Major Depressive Disorder, Bipolar Disorder, or Anxiety Disorder
20. Dementia Rating Scale < 135

Ages: 20 Years to 68 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 305 (Actual)
Dates: Start 2010-08; Primary Completion 2016-05 (Actual); Study Completion 2016-06-29 (Actual)

PRIMARY OUTCOMES:
Change from baseline in measures of executive control function and episodic memory at 6 months | 24 weeks
  tests of global intelligence, executive function, working memory and processing speed

SECONDARY OUTCOMES:
Change from baseline in brain structure, resting cerebral blood flow and network efficiency at 6 months | 24 weeks
  structural MRI (for gray matter density), resting CBF (cerebral blood flow, measured by arterial spin labeling) and cognitive activation fMRI studies
Change from baseline in measures of interleukin-6, tumor necrosis factor alpha, C-reactive protein at 6 months | Baseline and 24 weeks
Change from baseline in aerobic capacity at 6 months | 24 weeks
  aerobic capacity as measured by VO2 max
Change from baseline in measures of executive control function and episodic memory at 1 year | 48 weeks
  tests of global intelligence, executive function, working memory and processing speed

CONTACTS AND LOCATIONS:
Overall Officials: Richard P Sloan, PhD, Principal Investigator — Columbia University; Yaakov Stern, PhD, Principal Investigator — Columbia University
Locations (1):
- Richard Sloan, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Predovan D, Gazes Y, Lee S, Li P, Sloan RP, Stern Y. Effect of Aerobic Exercise on White Matter Tract Microstructure in Young and Middle-Aged Healthy Adults. Front Hum Neurosci. 2021 Jul 2;15:681634. doi: 10.3389/fnhum.2021.681634. eCollection 2021. PMID 34276329
- [Derived] Stern Y, MacKay-Brandt A, Lee S, McKinley P, McIntyre K, Razlighi Q, Agarunov E, Bartels M, Sloan RP. Effect of aerobic exercise on cognition in younger adults: A randomized clinical trial. Neurology. 2019 Feb 26;92(9):e905-e916. doi: 10.1212/WNL.0000000000007003. Epub 2019 Jan 30. PMID 30700591